CLINICAL TRIAL: NCT03031834
Title: Efficacy of Administration of Angiotensin Converting Enzyme Inhibition on Autonomic and Peripheral Neuropathy in Patients With Diabetes Mellitus
Brief Title: Efficacy of Administration of ACE-Inhibition on Autonomic and Peripheral Neuropathy in Patients With Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Konstantinos Tziomalos, Assistant Professor of Internal Medicine, Aristotle University Of Thessaloniki
Other Study IDs: AristotleUMEDSCH095
Record Dates: First submitted 2017-01-12; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Diabetic Autonomic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Quinapril

INTERVENTIONS:
Drug: Quinapril

SUMMARY:
Patients with diabetes mellitus and definite autonomic and peripheral neuropathy were randomized to receive quinapril or no treatment for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus with both autonomic and peripheral neuropathy

Exclusion Criteria:

* Hypertension, coronary heart disease

Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-01; Primary Completion 2001-05 (Actual)

PRIMARY OUTCOMES:
Changes in R-R variation during deep breathing | 2 years
Changes in response to Valsalva maneuver | 2 years
Changes in 30:15 ratio | 2 years
Changes in blood pressure response to standing | 2 years

IPD SHARING:
Plan to Share IPD: No